CLINICAL TRIAL: NCT06648590
Title: Pediococcus Acidilactici on Digestive Function and Well-being in Older Adults: a Randomized, Double-blind Placebo-controlled Trial
Brief Title: The Effect of Probiotics on the Improvement of Digestive Function and Well-being in the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wecare Probiotics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WK2024015
Record Dates: First submitted 2024-10-16; First posted 2024-10-18 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: People Aged 55-70 Years
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic grouptics (Experimental): 30B CFU/strip/day PA53, before meals; Storage:Store in a cool, dry place without sun exposure.
  Interventions: Dietary Supplement: Probiotic
- Placebo group (Placebo Comparator): Maltodextrin, one strip/day, before meals; Storage:Store in a cool, dry place without sun exposure.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — The experimental phase of this study lasts 56 days and each subject will have 3 follow-up visits(d1、d28、d56).
  Arms: Probiotic grouptics
Dietary Supplement: Placebo — The experimental phase of this study lasts 56 days and each subject will have 3 follow-up visits(d1、d28、d56).
  Arms: Placebo group

SUMMARY:
To evaluate the effectiveness and safety of the use of probiotics as food supplements compared to placebo in improving digestive function and well-being in older adults.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age is 55-70 years; 2) Willing to undergo 3 follow-up visits during the intervention period; 3) Willing to provide 2 blood, urine, and stool samples during the intervention period; 4) Willing to self-administer Pediococcus acidilactici PA53/placebo once daily during the intervention period; 5) Good eyesight, able to read and write, and can wear glasses; 6) Have good hearing and be able to hear and understand all instructions during the intervention.

Exclusion Criteria:

* 1) Suffering from digestive disorders, mainly gastrointestinal disorders (celiac disease, ulcerative colitis, Crohn's disease); 2) Has a severe neurological condition (epilepsy, stroke, severe head trauma, meningitis within the past 10 years, brain surgery, brain tumor, prolonged coma - excluding general anesthesia); 3) Has received/is receiving treatment for the following psychiatric disorders: alcohol/drug/substance abuse dependence, schizophrenia, psychosis, bipolar disorder; 4) Take medication for depression or low mood; 5) Suffering from internal organ failure (heart, liver, or kidney failure, etc.); 6) Radiotherapy or chemotherapy in the past; 7) Surgery/procedure under general anesthesia within the past three years, or planned to undergo a procedure/procedure under general anesthesia within the next 3 months during this trial; 8) Have had hepatitis (hepatitis B, hepatitis C), HIV or syphilis in the past; 9) Have taken Pediococcus acidilactici PA53 within the past 3 months.

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2024-10-20 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Change in GSRS scale | 56 days
  GSRS(Gastrointestinal Symptom Rating Scale) scale contains 13 items, each with 7 grades, from 0 to 6 indicating no symptoms, mild, mild, moderate, moderate-severe, severe, and very severe. A higher score on the GSRS scale indicates that the patient's gastrointestinal symptoms are more severe.

CONTACTS AND LOCATIONS:
Locations (1):
- Xu fei, Zhengzhou, Henan, China